CLINICAL TRIAL: NCT04403503
Title: The Influence of Tissue Adhesive to Palatal Donor Site Healing. A Randomized Controlled Clinical Trial
Brief Title: The Influence of Tissue Adhesive to Palatal Donor Site Healing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gencay Keceli, Assoc. Prof. Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Cyanoacrylate
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Donor Site Complication
MeSH Terms: interventions — Bucrylate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One author (H.G.K.) randomly assigned the patients, with 1:1 allocation ratio, into GS and GS+CY groups by making simple randomization without blocking (computer-generated randomization scheme) (Figure 1). Number-labeled opaque envelopes containing the name of assigned method were used for allocation concealment. The surgical procedures were carried out by (B.T.Y.) whereas another author (E.C.) acquired the intra- and post-operative data. No information regarding to the applied hemostatic was given to the patients to preserve the patient blinding.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gelatine Sponge (Active Comparator): After local anesthesia (2% articaine HCl with epinephrine 1:100,000) administration, palatal thickness was measured by perpendicularly inserting a Michigan-O periodontal probe from the corners of the rectangular donor area and mean value was recorded as 'palatal tissue thickness (PTT)'. Epithelialized gingival graft was harvested with the method described by Zucchelli et al.19 After a rectangular shaped initial incision, graft with 1-1.5 mm thickness was harvested approximately 1.5 to 3 mm away from gingival margins of upper teeth. After harvesting, excess fatty tissues were removed and de-epithelialization was performed to obtain DGG. Donor site was closed either with GS (Spongostan®, Ethicon, Somerville, USA)
  Interventions: Drug: Gelatin Sponge;Thrombin, Bovine 5000 IU Multiple Routes Kit [GELFOAM-JMI SPONGE KIT]
- Gelatine sponge +Cyanoacrylate (Active Comparator): After local anesthesia (2% articaine HCl with epinephrine 1:100,000) administration, palatal thickness was measured by perpendicularly inserting a Michigan-O periodontal probe from the corners of the rectangular donor area and mean value was recorded as 'palatal tissue thickness (PTT)'. Epithelialized gingival graft was harvested with the method described by Zucchelli et al.19 After a rectangular shaped initial incision, graft with 1-1.5 mm thickness was harvested approximately 1.5 to 3 mm away from gingival margins of upper teeth. After harvesting, excess fatty tissues were removed and de-epithelialization was performed to obtain DGG. Donor site was closed either with GS (Spongostan®, Ethicon, Somerville, USA) and GS covered with high viscosity CY (PeriAcryl®, Glustitch Inc., Delta, Canada) (GS+CY group)
  Interventions: Drug: Cyanoacrylate, Isobutyl

INTERVENTIONS:
Drug: Gelatin Sponge;Thrombin, Bovine 5000 IU Multiple Routes Kit [GELFOAM-JMI SPONGE KIT] — Donor site was closed either with GS (Spongostan®, Ethicon, Somerville, USA) (GS group)
  Arms: Gelatine Sponge
Drug: Cyanoacrylate, Isobutyl — Donor site was closed either with GS (Spongostan®, Ethicon, Somerville, USA) (GS group) and GS covered with high viscosity CY (PeriAcryl®, Glustitch Inc., Delta, Canada) (GS+CY group).
  Arms: Gelatine sponge +Cyanoacrylate

SUMMARY:
CTG was harvested from 21 patients in each group. Donor site was treated with either GS (control) or GS+CY (test). Palatal tissue thickness, graft dimensions, working time (WT) and primary bleeding time were recorded intraoperatively. The data of pain perception (PP) will be measured using visual analog scale, quantity of analgesics (QA), secondary bleeding (SB), epithelization level (EL), and color match (CM) will be assessed prospectively. these outcomes will be evaluated in the first 7 days and 14th, 21th, and 28th days. Patient reported outcomes will be recorded using OHIB 14 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18;
* PPS indication that needs CTG in anterior mandible;
* stable periodontium after phase I therapy;
* full-mouth plaque and bleeding scores <15%

Exclusion Criteria:

* previous palatal harvesting history;
* unstable endodontic conditions;
* tooth mobility at surgical site;
* systemic disease;
* pregnancy;
* use of medications with potential adverse effects to periodontal tissues

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Donor site pain perception (PP) | first week
  Patients score their daily donor site pain perception (PP) level by giving numbers from 0 to 10 according to the visual analog scale (VAS) (0: no pain, 1: minimal pain, 10: severe pain)

SECONDARY OUTCOMES:
Primary bleeding time (PBT) | during surgery
  Immediately after harvesting, sterile gauze was compressed to the palatal wound for 2 minutes, blood wiped once in every 30 seconds until bleeding stops. The duration was recorded as primary bleeding time (PBT).
Graft height (GH) | during surgery
  Dimensions were measured with periodontal probe
Graft width (GW) | during surgery
  Dimensions were measured with periodontal probe
Graft thickness (GT) | during surgery
  Dimensions were measured with periodontal probe
Working time (WT) | during surgery
  Harvesting process was recorded
Quantity of analgesics (QA) | first week
  Patients recorded the quantity of analgesics (QA) taken
Secondary bleeding (SB) | first week
  Patients recorded presence/absence of secondary bleeding (SB) (yes or no).
Sensation loss (SL) | first week, second week , third week, fourth week.
  Sensation loss (SL) was scored as none, medium or severe
Color match (CM) | first week, second week, third week, fourth week.
  Color match (CM) with the adjacent tissue was determined by using a VAS scale (0: absence of harmony, 10: excellent harmony)
Epithelization level (EL) | first week, second week, third week, fourth week.
  Epithelization level (EL) was scored as none, partial or full epithelization by means of bubble formation after dripping hydrogen peroxide (3%) to the wound surface following surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)